CLINICAL TRIAL: NCT03885960
Title: A Prospective Nationwide Study of Perthes' Disease in Norway: Functional and Radiographic Outcomes at a Mean Follow-up of Twenty Years
Brief Title: Perthes Disease in Norway
Status: Active, not recruiting | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: Sophies Minde Ortopedi (Industry)
Responsible Party: Principal Investigator, Stefan Huhnstock, Principal investigator, Oslo University Hospital
Other Study IDs: 2018/1924
Record Dates: First submitted 2019-01-09; First posted 2019-03-22 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Legg Calve Perthes Disease
Keywords: Hip; function; quality of life; osteoarthritis; Perthes; LCPD
MeSH Terms: conditions — Legg-Calve-Perthes Disease; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Calvé-Legg-Perthes disease (CLP) is a hip disease in children whose femoral head becomes completely or partially necrotic. The disease is most common in five-six years of age. The femoral head is gradually deformed during the active stages of the disease (5-7 years). By healing, the hip joint shape will vary from an approximately normal joint to pronounced changes, the hip joint will be irregular. Such a hip joint is available for osteoarthritis. The purpose of this study is to map the function of the hip, the patient's quality of life and especially the risk factors that affect the outcome of the previous CLP. A nationwide prospective study of CLP was conducted between 1996 and 2000. All children with newly diagnosed Perthes disease (425) were registered. The current study will follow up all these patients with an average follow-up of 20 years. Radiological endpoints are evidence of hip osteoarthritis. Patient-reported outcomes (PROMS) should illuminate the function of the hip and quality of life.

ELIGIBILITY:
Inclusion Criteria

- Subject was diagnosed with Perthes disease between 1996 and 2000 in Norway

Exclusion Criteria:

* Death upon follow up
* Other skeletal dysplasia
* Patient not able to give consent,

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients which have been diagnosed with Perthes disease in between 1996 and 2000 in Norway were registered and follow at least 5 years after diagnosis. All hospitals throughout Norway with orthopaedic service were included in the registration. Our study is a 20 years follow-up of the original study.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Hip osteoarthritis | an average of 20 years follow-up
  radiographic measurement of weight bearing zone
Hip function | an average of 20 years follow-up
  PROMS HOOS

SECONDARY OUTCOMES:
Hip ROM | an average of 20 years follow-up
  functional test of range of motion of the hip
Gluteal muscle strength | an average of 20 years follow-up
  Trendelenburg test
Hip strength | an average of 20 years follow-up
  single leg hop test - 6 meters

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Huhnstock, Phd, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital - Rikshospitalet, Oslo, Sognsvannsveien 20, Norway

DOCUMENTS (2):
  • Study Protocol (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT03885960/Prot_000.pdf
  • Informed Consent Form (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT03885960/ICF_001.pdf